CLINICAL TRIAL: NCT01657851
Title: An Open-Label, Randomized, Single Dose Crossover Study to Determine the Bioequivalence of Duodart® 0.5mg/0.4mg (Capsule Formulation of Dutasteride 0.5mg and Tamsulosin Hydrochloride 0.4mg) Compared to Concomitant Dosing of Avodart® 0.5mg and Omnic® 0.4mg Commercial Capsules in Healthy Male Subjects.
Brief Title: Bioequivalence - Duodart Against Avodart & Omnic
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 116502
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- dutasteride/tamsulosin (Experimental): The present study is planned to establish bioequivalence of Duodart® 0.5mg/0.4mg manufactured by GlaxoSmithKline to concomitant dosing with separate capsules of dutasteride 0.5 mg and tamsulosin hydrochloride 0.4 mg formulations commercially available in Russia.
  Interventions: Drug: dutasteride/tamsulosin
- dutasteride (Active Comparator): Dutasteride (Avodart®) is an approved potent dual type I and II, 5-alpha-reductase inhibitor indicated for the treatment of symptomatic benign prostatic hyperplasia (BPH) in men with an enlarged prostate to improve symptoms, reduce the risk of acute urinary retention and reduce the risk of the need for BPH-related surgery.
  Interventions: Drug: dutasteride; Drug: tamsulosin
- tamsulosin (Active Comparator): Tamsulosin (Omnic®) is an alpha-1A-adrenocepter blocking agent approved for the treatment of signs and symptoms of benign prostatic hyperplasia
  Interventions: Drug: dutasteride; Drug: tamsulosin

INTERVENTIONS:
Drug: dutasteride/tamsulosin — Duodart® 0.5 mg / 0.4 mg - 1 dose at Day 1 of each treatment period. There are 2 treatment periods separated by approximately a 28-day washout period. All study drugs will be administered orally as capsules
  Other Names: Duodart® 0.5 mg / 0.4 mg
  Arms: dutasteride/tamsulosin
Drug: dutasteride — Avodart® 0.5 mg together with Omnic® 0.4 mg - 1 dose at Day 1 of each treatment period. There are 2 treatment periods separated by approximately a 28-day washout period. All study drugs will be administered orally as capsules
  Other Names: Avodart® 0.5 mg
  Arms: dutasteride; tamsulosin
Drug: tamsulosin — Omnic® 0.4 mg together with Avodart® 0.5 mg - 1 dose at Day 1 of each treatment period. There are 2 treatment periods separated by approximately a 28-day washout period. All study drugs will be administered orally as capsules
  Other Names: Omnic® 0.4 mg
  Arms: dutasteride; tamsulosin

SUMMARY:
Open-label, randomized, single dose, two-treatment, two-way crossover study

DETAILED DESCRIPTION:
The present study is planned to establish bioequivalence of Duodart® 0.5mg/0.4mg manufactured by GlaxoSmithKline to concomitant dosing with separate capsules of dutasteride 0.5 mg and tamsulosin hydrochloride 0.4 mg formulations commercially available in Russia. The design of the present study relies on data obtained in pivotal bioequivalence study and Russian guidance on high quality bioequivalence studies.

Summary of treatment groups Treatment Sequence Number of subjects

1. 18
2. 18 Total number of subjects 36 Eligible subjects will be admitted to the research unit one day prior to dosing (Day 0) and will remain as inpatients until approximately 72 hours after dosing. Subjects will undergo a washout period of approximately 28 days from each dose of study medication. During washout period subjects will be contacted via telephone within approximately 10-14 days after the dosing for the collection of information about adverse events and medications taken by volunteers during washout period Overall study duration could be about 2 months - Screening up to 21 days + 10 days (5 days of each of 2 treatment periods) + 28 days washout period between treatment administration + 10-14 days of follow up period.

Upon completion of the last dosing session, subjects will be contacted via telephone within approximately 10-14 days for a follow-up inquiry (or visit at the discretion of the investigator) and will be subsequently discharged from the study.

* Order of Assessments and Procedures

Where multiple measurements/evaluations are scheduled for the same time then the measurements/evaluations will be taken in the following order:

1. Vital Signs
2. Orthostatic Vital Signs
3. PK - Blood Sample Where multiple measurements/evaluations are scheduled for the same time then the study co-coordinator will attempt to ensure that the PK samples are drawn as close to the scheduled time as possible whilst adhering to the order of assessments as described above.

   * Blinding and Randomisation On Day 0 of the first treatment period, subjects will be randomly allocated at the ratio of 1:1 to one of 2 treatments (refer to Table 1), according to a computer-generated randomisation list. CRO will generate the randomisation list. For the purpose of randomisation screening numbers of volunteers will be used; randomisation numbers will not be assigned to study subjects.

Treatment will be open-label; therefore, blinding procedures are not applicable.

* Number of Subjects Approximately 50 healthy male subjects will be screened to allow 36 eligible subjects to be randomized and ensure that 30 subjects complete the study according to the protocol without violations.
* PHARMACOKINETIC PARAMETERS
* Drug assay Dutasteride and tamsulosin will be extracted from human plasma by liquid-liquid extraction using organic solvent. Extracts will be analysed by validated high-performance liquid chromatography - mass spectrometry. The lower limit of detection is about 0.1ng/mL
* Calculation of Pharmacokinetic Parameters Pharmacokinetic parameters will be computed for each subject and treatment using standard methods as described in Appendix II.

For tamsulosin, the following PK parameters will be computed:

* Cmax
* Tmax
* AUC(0-t)
* AUC(0-∞)
* Half-life
* Mean residence time

For dutasteride, the following PK parameters will be computed:

* Cmax
* Tmax
* AUC(0-t)
* Mean residence time The half-life and AUC(0-∞) will be computed only for tamsulosin because duration of sampling period equal to 72 h is expected to be non-sufficient for reliable computation of half-life and AUC(0-∞) of dutasteride given the complex pharmacokinetics of dutasteride and long half-life of dutasteride at each of two elimination pathways [12].

  * ADVERSE EVENTS (AE) AND SERIOUS ADVERSE EVENTS (SAE) The investigator or site staff is responsible for detecting, documenting and reporting events that meet the definition of an AE or SAE.

AEs will be collected from the start of Study Treatment and until the follow-up contact.

SAEs will be collected over the same time period as stated above for AEs. However, any SAEs assessed as related to study participation (e.g. study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK product will be recorded from the time a subject consents to participate in the study up to and including any follow-up contact. All SAEs will be recorded and reported to GSK within 24 hours

* LIFESTYLE AND/OR DIETARY RESTRICTIONS
* Meals and meal composition Subjects will be required to fast for approximately 10 hours prior to dosing, with the exception of water, which will be allowed freely except for 1 hour before and 1 hour after dosing.

Following dosing, subjects will not be allowed food until 4 hours post dose. Meals will be served at the times outlined in Section 2 (Schedule of Assessments), in a seated position (unless orthostasis detected, in which meals should be served in a semi-recumbent position).

Meals will be served on Days 2 and 3 at approximately the same time as on Day 1.

Subjects will not be allowed to consume the following foods or drinks within 7 days prior to the first dose of study medication until after collection of the final pharmacokinetic blood sample: grapefruit juice; red wine; grapefruit or cruciferous vegetables (watercress, broccoli, cabbage, Brussels sprouts).

* Dosage and Administration One Duodart® 0.5mg/0.4mg capsule as Test formulation or one Avodart® 0.5 mg and one Omnic® 0.4 mg capsules as Reference formulation will be administered in the morning of Day 1 in each study period. The capsules should not be opened or chewed, but swallowed whole with 200 mL of water at room temperature
* STATISTICAL METHODS
* Population for analysis For pharmacokinetics parameters calculation and statistical analysis, the data received from no less than 30 volunteers who have completed the study according to the Protocol will be explored.

Safety analysis population of this study will consist of all volunteers who took part in at least one study stage.

Data from volunteers who discontinued the study prematurely will be included in the final report, but no included in the pharmacokinetics parameters calculation and statistical analysis.

If the volunteer has not taken any of the study drugs at all, his/her data are not to be included in the statistical analysis.

* Analysis Method For pharmacokinetics parameters calculation, statistical analysis, and results presentation statistical packages (Statistics, Microsoft Excel 2007, SAS, or SPSS) will be used.

Descriptive statistics will be used to present the mean value, standard deviation, median value, minimal and maximal value.

Analysis of variance will be done based on the assumption about the log-normal distribution of AUC, Cmax, and Cmax/AUC, and normal distribution of other pharmacokinetics parameters except tmax. The comparison of average values of the investigated and comparator drug parameters is performed with the multiplicative model as a basis and confidence intervals built for the ratio of the corresponding mean values. After the logarithmic transformation these values will be analyzed by analysis of variance (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent
* Males who are 18 - 45 years of age, inclusive
* Verified diagnosis "healthy"
* Body mass index 20-25 kg/m2 (inclusive)
* Negative results of test for HIV, syphilis, hepatitis B (HBs Ag) and hepatitis C
* Adequate, liver, and renal function
* adequate contraception

Exclusion Criteria:

* Poor metabolizer for CYP2D6
* Medical history of allergy
* Medical history of medicines intolerability
* Chronic diseases
* History of surgery on gastrointestinal tract
* History of prostate cancer
* History of breast cancer
* Acute infectious disease
* Regular use of drugs
* Intake of medicines with high influence on liver function or haemodynamics
* Use of drugs that influence activity of CYP2D6 and CYP3A4
* Use of Dutasteride less than 6 months before study entry or alpha-blockers less than 2 weeks before study entry
* Blood donation (≥450 mL of blood or plasma) less than 2 months before study start
* History of regular alcohol consumption
* A positive urine drug or alcohol
* Smoking more than 10 cigarettes a day
* Participation in Phase I clinical trials less than 3 months before study entry
* History of postural hypotension, dizziness, poor hydration, vertigo, vaso-vagal reactions or any other signs and symptoms of orthostasis
* Subjects who have consumed the following foods or drinks within 7 days prior to the first dose of study medication or at any time during the clinical phase of the study: grapefruit juice; red wine; grapefruit or cruciferous vegetables (watercress, broccoli, cabbage, Brussels sprouts).
* QTc ≥ 450 msec at screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2012-08-23 (Actual); Primary Completion 2012-12-05 (Actual); Study Completion 2012-12-05 (Actual)

PRIMARY OUTCOMES:
bioequivalence of a Combination Capsule formulation of dutasteride 0.5 mg/ tamsulosin HCl 0.4 mg (Duodart® 0.5 mg/ 0.4 mg fixed combination) relative to concomitant dosing of Avodart® 0.5 mg and the Omnic® 0.4 | 2 months
  Dutasteride and tamsulosin will be extracted from human plasma by liquid-liquid extraction using organic solvent. Extracts will be analysed by validated high-performance liquid chromatography - mass spectrometry. The lower limit of detection is about 0.1ng/mL

SECONDARY OUTCOMES:
to evaluate the safety and tolerability of the Combination Capsule formulation of dutasteride 0.5 mg/ tamsulosin HCl 0.4 mg | 2 months
  The following safety parameters will be assessed during the study: Physical examination; Orthostatic vital signs; Vital signs; 12-lead ECG; Adverse events; Serum chemistry; Complete blood count

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Reutov, Moscow Region, Russia

REFERENCES:
- See also: Results for study 116502 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116502?search=study&search_terms=116502#rs